CLINICAL TRIAL: NCT05609812
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Multicenter, Multinational Study to Evaluate the Efficacy and Safety of Atacicept in Subjects With Active Lupus Nephritis
Brief Title: Atacicept in Subjects With Active Lupus Nephritis (COMPASS)
Acronym: COMPASS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study recruitment is paused due to business reasons, but not due to regulatory or safety concerns.
Sponsor: Vera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VT-001-0070
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-10

CONDITIONS: Lupus Nephritis (LN)
Keywords: Systemic Lupus erythematosus (SLE); estimated glomerular filtration rate (eGFR); protenuria
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atacicept Dose (Experimental): Atacicept Dose once weekly subcutaneous (SC) Injection
  Interventions: Drug: Atacicept
- Placebo to match Atacicept (Placebo Comparator): Placebo to match Atacicept once weekly subcutaneous (SC) injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atacicept — Once weekly subcutaneous (SC) injections by prefilled syringe
  Other Names: VT-001
  Arms: Atacicept Dose
Drug: Placebo — placebo
  Arms: Placebo to match Atacicept

SUMMARY:
The objective of the study is to evaluate the effect of atacicept compared to placebo on changes to renal response in adult subjects with LN.

DETAILED DESCRIPTION:
The study will assess atacicept vs. placebo on the impact of renal function. Safety and patient reported outcomes will be clinically assessed. The clinical study is comprised of a 104 week double-blind treatment period, followed by a 52 week open-label treatment period and a 26 week safety follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or Female at least 18 years of age at time of signing consent
2. Must have the ability to understand and sign and date a written informed consent form
3. Diagnosis of SLE
4. Biopsy- Proven Active LN
5. Requires high-dose corticosteroids and immunosuppressive therapy for the treatment of active LN
6. Subject is willing to take oral MMF for the duration of the study

Key Exclusion Criteria:

1. eGFR of ≤30 mL/min/1.73 m2.
2. Sclerosis in 50% of glomeruli on renal biopsy.
3. Evidence of rapidly progressive glomerulonephritis.
4. Currently requiring renal dialysis or expected to require dialysis during the study.
5. Serum igG <7 g/L
6. Active infection or high infectious risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Renal Response as definedas UPCR ≤0.5 mg/mg, and eGFR ≥60 mL/min/1.73 m^2 or eGFR <60 mL/min/1.73 m^2 with no confirmed decrease from baseline of >20% | Week 52

SECONDARY OUTCOMES:
Renal Response with alternative success criteria | Weeks 52 and 104
Time to UPCR of≤0.5 mg/mg | Week 52
Renal Response at Week 104 | Week 104
Time to Death or Renal-Related Event | Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Curley, Study Director — Chief Development Officer
Locations (33):
- United States (26):
  - Vera Site # 0139, Huntsville, Alabama
  - Vera Site # 0138, La Jolla, California
  - Vera Site # 0127, La Palma, California
  - Vera Site # 0129, Long Beach, California
  - Vera Site # 0135, Northridge, California
  - Vera Site # 0136, Northridge, California
  - Vera Site # 0130, Santa Clarita, California
  - Vera Site # 0131, Torrance, California
  - Vera Site # 0143, New Haven, Connecticut
  - Vera Site # 0140, Gainesville, Florida
  - Vera Site # 0128, Miami, Florida
  - Vera Site # 0134, Atlanta, Georgia
  - Vera Site # 0137, Augusta, Georgia
  - Vera Site # 0144, Augusta, Georgia
  - Vera Site # 0147, Lawrenceville, Georgia
  - Vera Site # 0109, Chicago, Illinois
  - Vera Site # 0133, Las Vegas, Nevada
  - Vera Site # 0149, Summit, New Jersey
  - Vera Site # 0146, New York, New York
  - Vera Site # 0142, New York, New York
  - Vera Site # 0148, Cleveland, Ohio
  - Vera Site # 0145, Columbus, Ohio
  - Vera SIte # 0132, Jackson, Tennessee
  - Vera Site # 0125, Dallas, Texas
  - Vera Site # 0126, Dallas, Texas
  - Vera Site # 0122, El Paso, Texas
- Vera Site # 0141, Coto Laurel, Puerto Rico
- Spain (6):
  - Vera Site # 0349, A Coruña
  - Vera Site # 0348, Barcelona
  - Vera Site # 0347, Barcelona
  - Vera Site #0351, Santander
  - Vera Site # 0350, Seville
  - Vera Site # 0346, Valencia

REFERENCES:
- See also: Vera Therapeutics, Inc. Company Website — http://veratx.com